CLINICAL TRIAL: NCT03616873
Title: Early Mobilization of Older Adults in the Cardiovascular Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Lady Davis Institute (Other)
Collaborators: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Michael Goldfarb, Attending Staff, Division of Cardiology, Lady Davis Institute
Other Study IDs: 17-188
Record Dates: First submitted 2018-01-04; First posted 2018-08-06 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Physical Activity; Older Adults; Cardiovascular Diseases
MeSH Terms: conditions — Motor Activity; Cardiovascular Diseases | interventions — Early Ambulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults aged 60 or older
  Interventions: Other: Early Mobilization

INTERVENTIONS:
Other: Early Mobilization — The EM program consists of a progression of functional activities from level of function (LOF) 0 (lowest mobility) to 5 (highest mobility). Each LOF has 3 primary activities designed to promote the patient to the next level. The nurse will begin with mobility activities based on the LOF that matches the patient's current status. The nurse and clinical partner will attempt and/or complete each LOF activity once per shift.

SUMMARY:
An early mobilization (EM) program will be implemented in the Cardiovascular Intensive Care Unit at the Jewish General Hospital (JGH), an academic tertiary hospital in Montreal, Quebec.

The investigators will perform a prospective, pre/post-EM intervention study in adults aged ≥60 years old admitted to the Cardiovascular Intensive Care Unit (CICU) at the JGH. During a 3-month period, the investigators will prospectively enrol patients to the pre-intervention cohort. The EM intervention will then be implemented. During a 12-month period, the investigators will prospectively enrol patients to the intervention cohort. 1 and 12 months following hospital discharge, patients in the pre-intervention and post-intervention cohorts will be contacted by phone by a member of the research team to assess for functional status and quality of life measures.

The primary effectiveness outcome will be the mean improvement in level of function (LOF) during CICU admission and at 1 and 12 months. Covariates predicting improvement in LOF ("responsiveness") and ones which do not ("non-responsiveness") will be assessed. The recovery of physical function at 1 month and 6 months as measured by the SF-36 physical component summary score will be assessed. The SF-36 scores of the highest scoring tertile of LOF on hospital discharge will be compared with the lowest scoring tertile. Hospital readmission at 30 days and discharge home vs. healthcare facility will also be compared. For safety, the composite and individual components of the number of falls, injuries, and dislodgements over the total number of attempted mobility activities will be recorded. The results from the intervention cohort will be compared to the pre-intervention cohort for all results.

ELIGIBILITY:
Inclusion Criteria:

* Participating in early mobilization program
* Age 60 years old or older

Exclusion Criteria:

* CICU stays less than 24 hours
* Patients with prehospital LOF 0 (immobile), LOF 1 (bedbound) or 2 (can sit in chair only).
* Cardiac surgery patients will also be excluded.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the CICU in the early mobilization program aged 60 or older.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Mean change in Level of Function (LOF) scale score during CICU admission and 1 and 12 months post-hospitalization | Duration of Cardiac Intensive Care Unit stay (average 4 days) and 1 and 12 months post-hosptialization
  The mean improvement change in the Level of Function scale score in patients undergoing early mobilization. The Level of Function scale measures mobility and ranges from 0 (bed immobile) to 5 (walking more than 20 meters), with higher scores indicating better mobility.

SECONDARY OUTCOMES:
Recovery of physical function | 1 month and 12 months.
  Recovery of physical function at 1 month and 12 months as measured by the Short Form (SF)-36 physical component summary score (measures 8 subscales: physical functioning, physical role, bodily pain, general health, vitality, social functioning, emotional role and mental health). The score range is from 0 to 100 and scores are calibrated so that 50 is the average score. Higher scores mean less disability.
Recovery of functional ability | 1 month and 12 months
  The recovery of functional ability at 1 month and 12 months as measured by the Level of Function scale score. The Level of Function scale measures mobility and ranges from 0 (bed immobile) to 5 (walking more than 20 meters), with higher scores indicating better mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Goldfarb, MD, Principal Investigator — Lady Davis Institute
Locations (1):
- Jewish General Hospital / Lady Davis Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/73/NCT03616873/Prot_SAP_002.pdf
  • Informed Consent Form (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/73/NCT03616873/ICF_003.pdf